CLINICAL TRIAL: NCT03444181
Title: ALzheimer and MUsic THerapy: Effects of Music Lessons on Brain Plasticity, Mood, and Quality of Life in Alzheimer Patients
Acronym: ALMUTH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: NORCE Norwegian Research Centre AS (Other); Bergen Municipality (Unknown)
Responsible Party: Principal Investigator, Stefan Koelsch, Professor, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCN 260576
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; MCI With Increased Risk for Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music lessons (Experimental)
  Interventions: Behavioral: Music lessons
- Training intervention (Active Comparator)
  Interventions: Behavioral: Training intervention
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Music lessons — Also described as neurocognitive music therapy. Singing lessons will be provided once a week for a period of 12 months by a person with a qualification in music therapy, or by a person with a different relevant qualification (e.g. psychology and music teaching) under the supervision of a music therapist. Additionally, participants will have the opportunity to meet regularly (1-2 times per month) as a choir to sing the song they have learned together in a group.
  Arms: Music lessons
Behavioral: Training intervention — Cognitive training that is comparable in scope and extent to the music lessons, but not using music. Group training sessions will be provided once a week for a period of 12 months by a person with a qualification in physiotherapy or occupational therapy. Group activities may include group tours such as mountain hikes and the like (about 2 times per month) and will follow an established program for the elderly.
  Arms: Training intervention

SUMMARY:
Music has powerful effects on memory in patients with neurodegenerative diseases. However, although there is anecdotal evidence for beneficial effects of active music interventions in patients with Alzheimer's disease (AD), there is lack of high-quality research investigating this issue, and the cognitive, emotional, and social factors that contribute to potentially beneficial effects of music making in AD patients are largely unknown. In a randomised controlled intervention trial, a cohort of AD patients will undergo twelve months of music lessons specifically tailored for AD patients. Structural and functional magnetic resonance imaging (MRI) will be used to determine changes in brain age (as compared to two control groups), and voxel-based morphometry will be computed to determine contributions of different factors of the music intervention (cognitive, emotional, and social) to plastic changes of brain morphology, and a potential deceleration of brain atrophy. In addition, quality of life of patients. In cooperation with the Bergen municipality, and a strong network of national and international partners, the neurocognitive music therapy will be implemented, involving training of music therapists, and communication of results to patients, patient groups, and therapists.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer Disease
* Living independently at home (not in a care home or similar aged care facility)
* Able to complete questionnaires in Norwegian
* Able to undergo MRI scans
* Able to attend interventions and assessments in the area of Bergen, Norway
* Has given informed consent

Exclusion Criteria:

* Hearing impairment that cannot be mended by hearing aids
* Conditions that hinder MRI scans, such as claustrophobia or metal objects in body (e.g. pacemakers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2024-06-14 (Estimated); Study Completion 2024-06-14 (Estimated)

PRIMARY OUTCOMES:
Brain age | 12 months
  MRI-derived estimation of the deviation of a person's brain age from the chronological age of that same person, in months
Depression symptoms | 12 months
  Sum score of the Geriatric Depression Scale (GDS; 15 yes/no items; possible range of scores 0-15; higher scores indicating more severe depression symptoms)

SECONDARY OUTCOMES:
Living independently at home | 12 months and up to 5 years
  Whether a person still lives at home or has moved to a care home (time-to-event data)
Language abilities | 12 months
  Word Learning Test
Sensori-motor functions | 12 months
  Finger Tapping Test
Activities of daily living | 12 months
  Instrumental Activities of Daily Living (IADL)
Disease progression | 12 months
  Mini-Mental State Examination (MMSE)
Cognitive functioning | 12 months
  Stroop test, online version
Integrity of fibre tracts | 12 months
  Estimated from Diffusion Tensor Imaging (DTI)
Resting-state functional connectivity | 12 months
  Functional connectivity (posterior versus anterior/ventral) in default mode network (DMN)
Working alliance | 6 months
  Working Alliance Inventory-Short Revised (WAI-SR)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Koelsch, PhD, Principal Investigator — University of Bergen
Locations (1):
- Bergen Municipality, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Steen JT, van der Wouden JC, Methley AM, Smaling HJA, Vink AC, Bruinsma MS. Music-based therapeutic interventions for people with dementia. Cochrane Database Syst Rev. 2025 Mar 7;3(3):CD003477. doi: 10.1002/14651858.CD003477.pub5. PMID 40049590
- [Derived] Matziorinis AM, Flo BK, Skouras S, Dahle K, Henriksen A, Hausmann F, Sudmann TT, Gold C, Koelsch S. A 12-month randomised pilot trial of the Alzheimer's and music therapy study: a feasibility assessment of music therapy and physical activity in patients with mild-to-moderate Alzheimer's disease. Pilot Feasibility Stud. 2023 Apr 19;9(1):61. doi: 10.1186/s40814-023-01287-1. PMID 37076884
- [Derived] Flo BK, Matziorinis AM, Skouras S, Sudmann TT, Gold C, Koelsch S. Study protocol for the Alzheimer and music therapy study: An RCT to compare the efficacy of music therapy and physical activity on brain plasticity, depressive symptoms, and cognitive decline, in a population with and at risk for Alzheimer's disease. PLoS One. 2022 Jun 30;17(6):e0270682. doi: 10.1371/journal.pone.0270682. eCollection 2022. PMID 35771851
- See also: Project website — http://www.uib.no/en/brainandmusic/112850/alzheimer-and-music